CLINICAL TRIAL: NCT05206006
Title: Impact of Computerized Decision Support for ANTIBIOtic Prescription in Cancer Patients With Febrile NEutropenia in the Emergency Department on Treatment Failure. A Randomized Cluster-controlled Trial.
Brief Title: Impact of Computerized Decision Support for ANTIBIOtic Prescription in Cancer Patients With Febrile NEutropenia in the Emergency Department on Treatment Failure.
Acronym: ANTIBIONEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: APHP210357
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: Stepped wedged design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): As routine care, the choice of the initial antibiotic regimen will be let to the discretion of the emergency physician.
  Interventions: Other: routine care
- computerized decision support app (CDSA) Group (Experimental)
  Interventions: Other: Computerized Decision support app (CDSA)

INTERVENTIONS:
Other: routine care — The choice of the initial antibiotic regimen will be let to the discretion of the emergency physician
  Arms: Control Group
Other: Computerized Decision support app (CDSA) — Implementation of an Computerized Decision support app (CDSA) : physician will use this app to help him in the antibiotic choice. This app is an interactive algorithm based on international guidelines that takes into account patients' medical history and characteristics. Secondly, the application is also designed to propose an algorithm of antibiotic revaluation at day 3 for hospitalized patients, depending on patient clinical course, and biological and microbiological results. The revaluation suggests antimicrobial modification (escalation or de-escalation) or discontinuation and stopping rules with recommended duration of therapy also based on international guidelines.
  Arms: computerized decision support app (CDSA) Group

SUMMARY:
Treatment of patients with febrile neutropenia (FN) attending Emergency Departments (EDs) relies on rapid antibiotic initiation in order to control a presumed infection. The choice of initial antibiotics is empirical and depends on patient's prior colonization or infection by multi-drug resistant pathogens (MDRPs) and risk stratification. Stratification of high-risk patients needing broad-spectrum antibiotics is debated. Thus, for non-specialist physicians, this choice may be challenging, leading to inappropriate initial antimicrobial regimens, potential risks for the patient and higher costs. Furthermore, international guidelines recommended to develop antibiotic stewardship programs and promoted an initial strategy based on escalation or de-escalation approaches, with early reassessment depending on patients' clinical course and microbiological results. Nevertheless, this interesting strategy may increase the level of complexity for the choice of the initial antibiotic regimen by non-specialist emergency physicians who are often the first prescribers in this context.

We developed an interactive computerized decision support app (CDSA) for initial antibiotic prescription and early revaluation in patients with FN. The first goal of this app is to assist non-specialized physicians in choosing initial antimicrobial regimen for patients with FN when they attend EDs. It uses an interactive algorithm based on international guidelines that takes into account patients' medical history and characteristics. Secondly, the app is also designed to propose an algorithm of antibiotic revaluation at day 3-4 for hospitalized patients, depending on patient clinical course, and biological and microbiological results. The revaluation suggests antimicrobial modification (escalation or de-escalation) or discontinuation and stopping rules with recommended duration of therapy also based on international guidelines.

We hypothesize that such a CDSA may improve the adherence to guidelines for the choice of initial antibiotic regimen for FN in the ED, favour early antibiotic reassessment for hospitalized patients, both decreasing the risk of treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* reported or observed fever at arrival at the ED (≥38.3° C on one occasion or ≥38°C on two or more occasions within 1 h);
* chemotherapy-induced neutropenia (absolute neutrophil count ≤500/mm3 or ≤1000/mm3 and anticipated to decrease to fewer than 500/mm3 within 24 to 48 h).

Exclusion Criteria:

* refusal to participate;
* prior inclusion in the study for a previous episode of FN;
* any intravenous antibiotic administration during the preceding 72 h;
* renal failure requiring renal replacement therapy or with an estimated creatinine clearance of less than 20 ml/min;
* palliative status with life expectancy of less than three days;
* pregnancy, absence of health insurance, mental deficiency or inability to understand informed consent, no French speaking;
* patient with a microbiological documented infection when arriving at the ED (e.g. positive blood culture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2022-02-14 (Estimated); Primary Completion 2023-03-21 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 7 days following inclusion
  Treatment failure will be defined by any escalation of the assigned empirical initial antibiotic treatment (e.g. adjunction of aminoglycoside, glycopeptide or other anti-gram positive or any broadening of the beta-lactam spectrum) during the 7 days following inclusion, in relation with at least one of the following reasons:
  * microbiologic reason;
  * clinical progression of the presumed infection defined as persistence, recurrence or worsening of clinical signs or symptoms of presenting infection (e.g. death due to the initial infection, occurrence of sepsis or septic shock, need for oxygen therapy (or increasing oxygen flow) or mechanical or non-invasive ventilation in case of pneumonia, neurological deterioration in case of central nervous system infection). Treatment failure outcome will be reviewed by at least 2 experts blinded to the arm.

SECONDARY OUTCOMES:
Number of initial antibiotic regimen adhering to the international guidelines | at inclusion
Time to antibiotic initiation from patient triage at the emergency department (minutes) | at inclusion
Number of revaluations of initial antibiotic regimen at day 3 depending on patient clinical course and microbiological results; | at 3 days
Number of antimicrobial spectrum reductions | at 3 days
Number of antibiotic regimens with carbapenems, aminoglycosides or glycopeptides | at inclusion
Number of days of Carbapenems, aminoglycosides and glycopeptides therapy | up to 3 months
Number of super-infections | up to 3 months
  A super-infection will be defined as new, persistent or worsening symptoms and/or signs of infection associated with the isolation of a new pathogen (different, or different susceptibilities) or the development of a new site of infection;
Number of super-infections due to clostridium difficile | up to 3 months
Number of colonization | up to 3 months
  Colonization will be defined as isolation during or after therapy of Gram-negative bacteria resistant to the beta-lactam included in the empirical regimen, without symptoms or signs of infection
Number of episodes of nephrotoxicity | up to 3 months
Number of episodes of other toxicities | up to 3 months
  Toxicities will be defined according to the common terminology criteria for adverse events
Occurrence of any complication during hospital stay or follow-up | up to 3 months
Number of re-hospitalizations due to a complication related to the initial infection | within 7 days of discharge
Antibiotic treatment duration | up to 3 months
Length of hospital stay | up to 3 months
Total 3-month costs | at 3 months
Number of deaths related to infection | at 3 months
  Death related to infections will be defined according to the physician in charge of the patient
Number of in-hospital death | up to 3 months
Survival status | at day 90
Health related quality of life | at inclusion
  Quality of life will be assessed using the EQ5D5L scale. The EQ5D5L scale is composed of two parts: a descriptive system and the EQ Visual Analog Scale (EQ VAS). The descriptive system has five dimensions. Each dimension has five levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The descriptive system ranges from 1 to 25, the higher the score the worse the quality of life. The score goes from VAS 0 to 100, the higher the VAS score the better the quality of life.
Health related quality of life. | at day 30
  Quality of life will be assessed using the EQ5D5L scale. The EQ5D5L scale is composed of two parts: a descriptive system and the EQ Visual Analog Scale (EQ VAS). The descriptive system has five dimensions. Each dimension has five levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The descriptive system ranges from 1 to 25, the higher the score the worse the quality of life. The score goes from VAS 0 to 100, the higher the VAS score the better the quality of life.
Health related quality of life. | at 3 months
  Quality of life will be assessed using the EQ5D5L scale. The EQ5D5L scale is composed of two parts: a descriptive system and the EQ Visual Analog Scale (EQ VAS). The descriptive system has five dimensions. Each dimension has five levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The descriptive system ranges from 1 to 25, the higher the score the worse the quality of life. The score goes from VAS 0 to 100, the higher the VAS score the better the quality of life.

IPD SHARING:
Plan to Share IPD: Undecided